CLINICAL TRIAL: NCT00336583
Title: Phase II Study of Etoposide, Methylprednisolone, High-dose Cytarabine and Oxaliplatin (ESHAOX) for Patients With Refractory or Relapsed Non-Hodgkin's Lymphoma
Brief Title: Etoposide, Methylprednisolone, High-dose Cytarabine and Oxaliplatin as 2nd Line Therapy for Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Suh, Cheolwon, AsanMedical Center, University of Ulsan College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC 2006-130
Record Dates: First submitted 2006-06-13; First posted 2006-06-14 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2009-09

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: oxaliplatin; ESHAOX; refractory; relapsed; non-hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — Oxaliplatin; Etoposide; Methylprednisolone; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxaliplatin, response (Experimental): relapsed or refractory non-Hodgkin's lymphoma
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin, 130 mg per square meter, on day 1
  Other Names: etoposide, 40 mg per square meter on days 1 to 4,; methylprednisolone, 500 mg on days 1 to 5,; cytarabine, 2 g per square meter on day 5

SUMMARY:
Oxaliplatin will be used instead of cisplatin in well-known salvage regimen of etoposide, methylprednisolone, cytarabine and cisplatin (ESHAP). Clinical efficacy and toxicity of this ESHAOX salvage regimen will be evaluated in refractory or relapsed non-Hodgkin's lymphoma patients.

DETAILED DESCRIPTION:
Patients with aggressive non-Hodgkin's lymphoma (NHL) are known to have a malignancy considered curable in many cases. However, diagnosis of refractory or relapsed disease is devastating and the treatment is difficult because regimens of chemotherapy used as salvage therapy are available only in limited numbers. ESHAP, consisting of etoposide, methylprednisolone, high-dose cytarabine and cisplatin, is one of commonly used salvage regimen, and showed its efficacy and feasibility. But it often requires discontinuation of the treatment due to its myelosuppression, neuropathy and renal toxicity, which can also impede further treatment. Oxaliplatin, a platinum coordination complex with an oxalato-ligand as the leaving group and a 1,2-diaminocyclohexane carrier, possesses higher cytotoxic potency on molar basis than cisplatin and carboplatin, and was reported to be active in patients with NHL as a single agent. In addition, the substitution of cisplatin by oxaliplatin in the DHAP regimen, another commonly used one in relapsed or refractory NHL, showed meaningful anti-tumor activity with favorable toxicity profile. Based on preclinical and clinical findings, we will conduct a multi-center phase II study of ESHAOX, which substitutes oxaliplatin with cisplatin in the ESHAP regimen, to evaluate the efficacy and toxicity profile in patients with recurrent or refractory NHL.

ELIGIBILITY:
Inclusion Criteria:

* Previously histologically confirmed aggressive lymphomas, defined according to WHO classification (except Burkitt's lymphoma, lymphoblastic lymphoma)
* Failure to achieve a complete remission with the initial induction chemotherapy, or recurrent disease
* Performance status (ECOG) ≤3
* Age ≤ 75
* Treated with at least one CHOP or CHOP-derived doxorubicin containing regimen
* At least one or more uni-dimensionally measurable lesion(s) defined as; ≥2 cm by conventional CT or ≥ 1 cm by spiral CT or skin lesion (photographs should be taken) or measurable lesion by physical examination
* Adequate organ functions defined as; ANC > 1,500/ul, platelet > 75,000/ul, transaminases < 3 X upper normal values; bilirubin < 2 mg%
* Written informed consent approved by Institutional Review Board

Exclusion Criteria:

* Any other malignancies within the past 5 years except skin basal cell ca or CIS of cervix
* Serious co-morbid diseases
* Pregnancy or breast-feeding

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-06; Primary Completion 2006-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheolwon Suh, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Sym SJ, Lee DH, Kang HJ, Nam SH, Kim HY, Kim SJ, Eom HS, Kim WS, Suh C. A multicenter phase II trial of etoposide, methylprednisolone, high-dose cytarabine, and oxaliplatin for patients with primary refractory/relapsed aggressive non-Hodgkin's lymphoma. Cancer Chemother Pharmacol. 2009 Jun;64(1):27-33. doi: 10.1007/s00280-008-0847-y. Epub 2008 Oct 7. PMID 18839172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 27 patients were enrolled between April and December 2006 from eight institutions in South Korea.
Pre-assignment Details: Patients with symptomatic central nervous system involvement and pregnant or breastfeeding women were excluded. Patients with grade 2 or more peripheral neuropathy at the time of study entry were also excluded.
Groups:
- ESHAOx: The ESHAOx consisted of Etoposide (40 mg per square meter on days 1-4), Methylprednisolone (500 mg on days 1-5), Cytarabine (2 g per square meter on day 5), and Oxaliplatin (130 mg per square meter on day 1) every 3 weeks to a maximum of six cycles.
Period: Overall Study
Arm/Group | ESHAOx
Started | 27
Completed | 25
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | ESHAOx
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 17
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 27

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The Overall Response Rate was measured by the number of patients per the total treatment population who partially or completely responded to treatment. Response was evaluated according to the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas.
Time Frame: up to 24 weeks
Population: 25 patients who had completed at least 3 cycles of ESHAOx study treatment were analyzed. 2 patients who did not complete 3 cycles of study treatment were excluded from the response analysis.
Measure: Number; unit: pariticipants
Arm/Group | ESHAOx
Number analyzed (Participants) | 25
pariticipants | 17

2. Secondary Outcome: Worst Toxicity Grade by Patient
Description: graded by National Cancer Institute Common Toxicity Criteria of Adverse Event version 3.0
Time Frame: up to 24 weeks
Population: The 27 patients received a total of 103 cycles of the ESHAOx treatment, with a median number of four cycles per patient. Except one who was lost to follow-up after one cycle, 26 patients were assessable for toxicity.
Measure: Number; unit: participants
Arm/Group | ESHAOx
Number analyzed (Participants) | 26
participants
  Grade 1 neutropenia | 3
  Grade 2 neutropenia | 3
  Grade 3 neutropenia | 2
  Grade 4 neutropenia | 13
  Grade 1 thrombocytopenia | 4
  Grade 2 thrombocytopenia | 3
  Grade 3 thrombocytopenia | 3
  Grade 4 thrombocytopenia | 6

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | ESHAOx
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ESHAOx (N=26)
febrile neutropenia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ESHAOx (N=26)
neutropenia grade 1 (Blood and lymphatic system disorders) | 3 (3)
neutropenia grade 2 (Blood and lymphatic system disorders) | 3 (3)
neutropenia grade 3 (Blood and lymphatic system disorders) | 2 (2)
neutropenia grade 4 (Blood and lymphatic system disorders) | 13 (13)
thrombocytopenia grade 1 (Blood and lymphatic system disorders) | 4 (4)
thrombocytopenia grade 2 (Blood and lymphatic system disorders) | 3 (3)
thrombocytopenia grade 3 (Blood and lymphatic system disorders) | 3 (3)
thrombocytopenia grade 4 (Blood and lymphatic system disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes